CLINICAL TRIAL: NCT03705793
Title: Effectiveness of Mometasone Nasal Irrigation for Chronic Rhinosinusitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201801067
Record Dates: First submitted 2018-10-08; First posted 2018-10-15 (Actual); Results first posted 2020-12-19 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Chronic Rhinosinusitis (Diagnosis); Allergic Rhinosinusitis; Chronic Eosinophilic Rhinosinusitis
Keywords: mometasone irrigation chronic rhinosinusitis; mometasone spray; rhinosinusitis
MeSH Terms: conditions — Disease; Rhinitis, Allergic, Perennial; Rhinosinusitis | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mometasone Furoate Nasal Irrigation (Experimental): The study intervention will be mometasone furoate powder (1.2 mg/capsule) and placebo nasal spray. The placebo nasal spray will contain the same inert ingredients found in MF nasal spray: glycerin, microcrystalline cellulose and carboxymethylcellulose, sodium citrate, citric acid, benzalkonium chloride, and polysorbate 80. The placebo nasal spray will be packaged identically to the mometasone nasal spray. Participants will be required to dissolve the contents of two capsules into an 8-ounce (240 mL) sinus rinse bottle along with the saline rinse. All participants will be instructed to perform the following once daily: irrigation of both right and left nasal cavity with one-half of the contents of the nasal rinse followed by 2 sprays per nostril of the nasal spray.
  Interventions: Drug: Mometasone Furoate Nasal Irrigation
- Mometasone Nasal Spray (Active Comparator): The study intervention will be mometasone nasal spray (50 mcg/spray) and placebo nasal irrigation. The placebo will contain lactose monohydrate and will be supplied in capsules identical to the budesonide capsules. Participants will be required to dissolve the contents of the two capsules into an 8-ounce (240 mL) sinus rinse bottle along with the saline rinse. All participants will be instructed to perform the following once daily: irrigation of both right and left nasal cavity with one-half of the contents of the nasal rinse followed by 2 sprays per nostril of the nasal spray.
  Interventions: Drug: Mometasone Nasal Spray

INTERVENTIONS:
Drug: Mometasone Furoate Nasal Irrigation — Participants will undergo an 8-week treatment course that includes nasal saline irrigation with mometasone powder and placebo nasal spray.
  Arms: Mometasone Furoate Nasal Irrigation
Drug: Mometasone Nasal Spray — Participants will undergo an 8-week treatment course that includes placebo saline irrigation with mometasone nasal spray.
  Other Names: Nasonex
  Arms: Mometasone Nasal Spray

SUMMARY:
Chronic rhinosinusitis (CRS) affects up to 12.5% of the US population and has a significant disease burden. The recommended medical management of CRS includes large-volume, low-pressure saline lavage, systemic antibiotics, and intranasal corticosteroids (INCS). While the efficacy and safety of INCS are well-established for the long-term management of CRS, penetration of INCS beyond the nasal vestibule and into the paranasal sinuses is limited. The aim of this study is to evaluate the effectiveness of mometasone furoate large-volume, low-pressure nasal irrigation for surgery-naive CRS patients.

DETAILED DESCRIPTION:
Mometasone furoate nasal spray (MFNS) is a INCS that is used in the management of CRS. The overall goal of this proposed research project is to optimize topical delivery of MF to the paranasal sinuses in surgery-naive CRS patients through the use of high-volume, low-pressure nasal saline irrigation. The investigators will be conducting a single-site, double-blinded, placebo-controlled randomized clinical trial (RCT) in which we propose to evaluate the effectiveness of MF nasal irrigation compared to MF nasal spray.

ELIGIBILITY:
Inclusion Criteria:

12-weeks or longer of two or more of the following signs and symptom consistent with CRS:

* mucopurulent drainage(anterior, posterior, or both)
* nasal obstruction (congestion)
* facial pain-pressure-fullness
* and decreased sense of smell

AND inflammation documented by one or more of the following findings:

* purulent mucus or edema in the middle meatus or ethmoid region
* radiographic imaging showing inflammation of the paranasal sinuses.

Exclusion Criteria:

* inability to speak or understand English
* nasal polyps
* history of nasal or sinus surgery
* comorbid mucociliary conditions
* dependence on prolonged corticosteroid therapy for comorbid conditions, such as asthma and chronic obstructive pulmonary disease
* history of oral or systematic antibiotic use in the past 2 weeks
* history of allergy to MF or other topical steroids
* pregnant or breastfeeding
* participants with a baseline SNOT-22 score of 9 or less will be excluded due to inability to achieve a minimally clinically improved difference pre- and post-intervention.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Washington University, St Louis, Missouri

REFERENCES:
- [Background] Meltzer EO, Hamilos DL, Hadley JA, Lanza DC, Marple BF, Nicklas RA, Bachert C, Baraniuk J, Baroody FM, Benninger MS, Brook I, Chowdhury BA, Druce HM, Durham S, Ferguson B, Gwaltney JM Jr, Kaliner M, Kennedy DW, Lund V, Naclerio R, Pawankar R, Piccirillo JF, Rohane P, Simon R, Slavin RG, Togias A, Wald ER, Zinreich SJ; American Academy of Allergy, Asthma and Immunology; American Academy of Otolaryngic Allergy; American Academy of Otolaryngology-Head and Neck Surgery; American College of Allergy, Asthma and Immunology; American Rhinologic Society. Rhinosinusitis: Establishing definitions for clinical research and patient care. Otolaryngol Head Neck Surg. 2004 Dec;131(6 Suppl):S1-62. doi: 10.1016/j.otohns.2004.09.067. PMID 15577816
- [Background] Ray NF, Baraniuk JN, Thamer M, Rinehart CS, Gergen PJ, Kaliner M, Josephs S, Pung YH. Healthcare expenditures for sinusitis in 1996: contributions of asthma, rhinitis, and other airway disorders. J Allergy Clin Immunol. 1999 Mar;103(3 Pt 1):408-14. doi: 10.1016/s0091-6749(99)70464-1. PMID 10069873
- [Background] Bhattacharyya N, Orlandi RR, Grebner J, Martinson M. Cost burden of chronic rhinosinusitis: a claims-based study. Otolaryngol Head Neck Surg. 2011 Mar;144(3):440-5. doi: 10.1177/0194599810391852. Epub 2011 Feb 3. PMID 21493210
- [Background] Kalish LH, Arendts G, Sacks R, Craig JC. Topical steroids in chronic rhinosinusitis without polyps: a systematic review and meta-analysis. Otolaryngol Head Neck Surg. 2009 Dec;141(6):674-83. doi: 10.1016/j.otohns.2009.08.006. PMID 19932837
- [Background] Rudmik L, Hoy M, Schlosser RJ, Harvey RJ, Welch KC, Lund V, Smith TL. Topical therapies in the management of chronic rhinosinusitis: an evidence-based review with recommendations. Int Forum Allergy Rhinol. 2013 Apr;3(4):281-98. doi: 10.1002/alr.21096. Epub 2012 Oct 8. PMID 23044832
- [Background] Thomas WW 3rd, Harvey RJ, Rudmik L, Hwang PH, Schlosser RJ. Distribution of topical agents to the paranasal sinuses: an evidence-based review with recommendations. Int Forum Allergy Rhinol. 2013 Sep;3(9):691-703. doi: 10.1002/alr.21172. Epub 2013 May 31. PMID 23729216
- [Background] Harvey RJ, Schlosser RJ. Local drug delivery. Otolaryngol Clin North Am. 2009 Oct;42(5):829-45, ix. doi: 10.1016/j.otc.2009.07.005. PMID 19909862
- [Background] Snidvongs K, Pratt E, Chin D, Sacks R, Earls P, Harvey RJ. Corticosteroid nasal irrigations after endoscopic sinus surgery in the management of chronic rhinosinusitis. Int Forum Allergy Rhinol. 2012 Sep-Oct;2(5):415-21. doi: 10.1002/alr.21047. Epub 2012 May 7. PMID 22566474
- [Background] Bachert C, Meltzer EO. Effect of mometasone furoate nasal spray on quality of life of patients with acute rhinosinusitis. Rhinology. 2007 Sep;45(3):190-6. PMID 17956016
- [Background] Mosges R, Bachert C, Rudack C, Hauswald B, Klimek L, Spaeth J, Rasp G, Vent J, Hormann K. Efficacy and safety of mometasone furoate nasal spray in the treatment of chronic rhinosinusitis. Adv Ther. 2011 Mar;28(3):238-49. doi: 10.1007/s12325-010-0105-7. Epub 2011 Feb 3. PMID 21318604
- [Background] Derendorf H, Meltzer EO. Molecular and clinical pharmacology of intranasal corticosteroids: clinical and therapeutic implications. Allergy. 2008 Oct;63(10):1292-300. doi: 10.1111/j.1398-9995.2008.01750.x. PMID 18782107

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Mometasone Furoate Nasal Irrigation Arm 3 participants lost to follow-up 2 participants withdrew
  Mometasone Nasal Spray Arm 4 participants lost to follow-up
  1 participant withdrew
  While 53 participants were initially enrolled, a total of 7 participants were lost to follow-up and 3 participants withdrew. Thus, the total number of participants who completed the study was 43.
Period: Overall Study
Arm/Group | Mometasone Furoate Nasal Irrigation | Mometasone Nasal Spray
Started | 27 | 26
Completed | 22 | 21
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: An intention-to-treat approach was used for all data analyses, which included all patients who were enrolled and randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate Nasal Irrigation | Mometasone Nasal Spray | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Median (Full Range); unit: years] | 48 [19 to 67] | 50 [19 to 66] | 48 [19 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 11 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 17 | 21 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Overall Comorbidity [Count of Participants; unit: Participants]
  None | 14 | 12 | 26
  Mild | 6 | 12 | 18
  Moderate | 2 | 3 | 5
  Severe | 4 | 0 | 4
Endoscopy Grading Scale [Median (Full Range); unit: units on a scale] — Nasal endoscopy score is derived from Lund Kennedy System for polyps , discharge, and edema on a scale of 0-12 with higher values indicating worse outcome.
  Polyps graded from 0 to 2 (0=absent, 1=limited to middle meatus, 2=extending to nasal cavity) Discharge graded from 0 to 2 (0=absent, 1=thin/clear, 2=thick) Edema graded from 0 to 2 (0=absent, 1=mild/moderate, 2=polypoid degeneration) VAS is graded patient's subjective perception of sense of smell with 0 indicating total anosmia and 5 normal olfaction.
  units on a scale | 4 [1 to 8] | 4 [0 to 8] | 4 [0 to 8]
SINO-NASAL OUTCOME TEST (SNOT-22) [Median (Full Range); unit: units on a scale] — Rating severity of a list of 22 items (symptoms and social/emotional consequences of rhinosinusitis) using a scale of 0 to 5; 0=No problem; 1=Very mild problem; 2=Mild or slight problem; 3=Moderate problem; 4=Severe problem; and 5=Problem as bad as it can be. Each of the 22 items is rated on a scale of 0 to 5 for min-max range of scores of 0 to 110
  units on a scale | 50 [12 to 99] | 40 [11 to 71] | 42 [11 to 99]

OUTCOME MEASURES:

1. Primary Outcome: Change in Sino-Nasal Outcome Test Scores (SNOT-22)
Description: The change in Sino-Nasal Outcome Test scores (SNOT-22) scores pre- and post-treatment between the two arms was measured. The Sino-Nasal Outcome Test asks subjects to rate how "bad" their rhinosinusitis is by using a 0-5 point scale with 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be. The SNOT includes 22 questions (symptoms and social/emotional consequences of rhinosinusitis), each of which are rated from 0 to 5 for a minimum score of 0 to maximum score of 110, with higher scores representing worse outcome.
  All relevant time points used in the calculation in the Time Frame (e.g., 'baseline and 8 weeks")
Time Frame: Change from Baseline to Week 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mometasone Furoate Nasal Irrigation | Mometasone Nasal Spray
Number analyzed (Participants) | 24 | 23
score on a scale | 23.18 [15.7 to 30.7] | 17.7 [10.3 to 25.04]

2. Secondary Outcome: Number of Participants Who Score <3 on the Clinical Global Impression Scale
Description: CGI asks subjects to rate their overall response to treatment using a 7-point Likert scale with anchors of 1=very much improved, 4=no change, and 7=very much worse.
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Mometasone Furoate Nasal Irrigation | Mometasone Nasal Spray
Number analyzed (Participants) | 24 | 23
Participants | 22 | 20

3. Secondary Outcome: Change in Nasal Endoscopic Findings Using the Lund-Kennedy Grading System
Description: A board-certified otolaryngologist will perform a nasal endoscopic examination pre- and post-intervention and findings recorded using the Lund-Kennedy grading system.
  The The Lund Kennedy System grades the pathologic state of the nasal cavity based on the presence of polyps, nasal discharge, and mucosal edema.
  Polyps graded from 0 to 2 (0=absent, 1=limited to middle meatus, 2=extending to nasal cavity) Discharge graded from 0 to 2 (0=absent, 1=thin/clear, 2=thick) Edema graded from 0 to 2 (0=absent, 1=mild/moderate, 2=polypoid degeneration). Scores are added for each side of the nose with a minimum score of 0 and maximum score of 12 with higher scores indicating more severe sinonasal inflammation.
Time Frame: Change from Baseline to Week 8
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mometasone Furoate Nasal Irrigation | Mometasone Nasal Spray
Number analyzed (Participants) | 24 | 23
units on a scale | 2.2 [1.1 to 3.3] | 2.1 [1.0 to 3.1]

ADVERSE EVENTS:
Time Frame: Up to 8 weeks. Adverse events were monitored/assessed through study completion.
Description: Number of participants at risk is based on the number of participants who were randomized and allocated to the 2 arms. The number stated in the participant flow is the number of participants who completed the trial.
Arm/Group | Mometasone Furoate Nasal Irrigation | Mometasone Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate Nasal Irrigation (N=26) | Mometasone Nasal Spray (N=27)
myocardial infarction (Cardiac disorders) | 0 | 1 (1) — 1 patient had a myocardial infarction during the study enrollment. However, the serious adverse event was not considered to be related to the study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT03705793/Prot_SAP_001.pdf